CLINICAL TRIAL: NCT03507582
Title: A Feasibility and Usability Study of a Nursing Orchestrated, Customized 3 Dimensional Virtual Reality Environment in Children With Hemophilia Undergoing Routine Intravenous Procedures
Brief Title: Virtual Reality for Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB16-00403
Record Dates: First submitted 2018-04-13; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Active Comparator): This intervention consists of a disposable virtual reality headset which will enable the use of virtual reality in clinic through the commodity hardware iPod Touch. An additional piece of software on an iPad will allow clinical staff to act as an orchestrator and trigger events that occur for the patient's benefit in the virtual reality environment. The mechanism for the dashboard will be dashboard software running on an iPad tablet that will wirelessly communicate to the iPod Touch the patient is wearing. A study timer will be incorporated into the orchestration dashboard. The VAS/FACES scale will be incorporated into the iPad used for orchestration.
  Interventions: Other: Virtual Reality Distraction
- Standard of Care Distraction (Active Comparator): This intervention consists of a two dimensional distraction (ie TV/tablet) as well as verbal distraction (ie singing/talking/music) will be allowed by caregivers, nurses and phlebotomy staff but will not qualified or quantified. IV procedures will proceed in Groups A and B. At the completion of the IV procedure the nurse orchestrator will stop the procedure timer. The Subject, Guardian and Nurse orchestrator will complete the Final VAS/FACES assessment on the iPad.
  Interventions: Other: Standard of Care Distraction

INTERVENTIONS:
Other: Virtual Reality Distraction — This intervention consists of a disposable virtual reality headset which will enable the use of virtual reality in clinic through the commodity hardware iPod Touch. An additional piece of software on an iPad will allow clinical staff to act as an orchestrator and trigger events that occur for the patient's benefit in the virtual reality environment. The mechanism for the dashboard will be dashboard software running on an iPad tablet that will wirelessly communicate to the iPod Touch the patient is wearing. A study timer will be incorporated into the orchestration dashboard. The VAS/FACES scale will be incorporated into the iPad used for orchestration.
  Arms: Virtual Reality Distraction
Other: Standard of Care Distraction — This intervention consists of a two dimensional distraction (ie TV/tablet) as well as verbal distraction (ie singing/talking/music) will be allowed by caregivers, nurses and phlebotomy staff but will not qualified or quantified. IV procedures will proceed in Groups A and B. At the completion of the IV procedure the nurse orchestrator will stop the procedure timer. The Subject, Guardian and Nurse orchestrator will complete the Final VAS/FACES assessment on the iPad.
  Arms: Standard of Care Distraction

SUMMARY:
Children with hemophilia are exposed to intravenous (IV) procedures that cause pain/anxiety and distraction methods can be employed to improve the patient experience. Three-dimensional virtual reality (VR) environments can reduce distress related to procedures. To be utilized in a clinical setting, however, these devices must address infection control concerns and fit pediatric patients. Additionally, for use in hemophilia care, environments should encourage a subject to keep their hands/arms still to facilitate procedures. Nursing orchestration of the VR environment via an iPad dashboard has the potential to increase feasibility and acceptance by patients, families and providers of the VR experience without disrupting routine clinical care.

DETAILED DESCRIPTION:
Patients with hemophilia A and B (HA/HB) are frequently treated with IV infusions of clotting factor concentrates to treat and prevent bleeding. Additionally they typically have at least yearly IV laboratory assessments. Pain and anxiety with needle related procedures particularly in children with hemophilia can lead to development of needle phobia, treatment avoidance and poor adherence to treatment regimens. Conventional virtual reality (VR) environments have been shown to reduce pain/anxiety in pediatric populations however in a clinical setting children with hemophilia have specific VR design needs that have not been addressed. Certain issues related to VR environments are related to the pediatric age range. These include the size and weight of VR headsets, the ease of donning and doffing headsets, and degree of engagement with VR environments. Hemophilia specific issues include the need for the VR experience to limit movement of the hands/arms to facilitate IV procedures, customization to prevent boredom/disengagement from repeated use and ability of clinical staff to trigger events via an orchestration dashboard that occur for the patients benefit at key times during IV procedures. Lastly, there are issues related to integration into a clinical setting. These include ability to integrate into clinical care without adversely affecting clinic flow, and infection control issues related to headset design.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent form
2. Willing to comply with all study procedures and be available for the duration of the study
3. Diagnosed with Hemophilia A or B
4. Male or female, aged >6 years to <19 years
5. Subject and caregiver able to understand and speak English
6. Being seen for routine comprehensive hemophilia care visits during which an IV procedure is planned as standard of care.

Exclusion Criteria:

1. Inability to use the VR equipment (ie visual, cognitive or hearing impairment that would preclude engagement with the VR environment)
2. History of motion sickness as reported by patient or caregiver
3. History of poorly controlled seizures as reported by patient or caregiver

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Nurse Orchestrated Virtual Reality Distraction | Twelve months
  The primary outcome of feasibility was assessed using a surrogate marker of feasibility which was duration of the IV procedure measured in minutes in both study arms. Procedure time was the length of time from the moment a patient was positioned for the procedure to the completion of the procedure. The study timer was incorporated in the study IPAD and timing was performed by the nurse orchestrator.
Standard of Care Distraction | Twelve months
  The primary outcome of feasibility was assessed using a surrogate marker of feasibility which was duration of the IV procedure measured in minutes in both study arms. Procedure time was the length of time from the moment a patient was positioned for the procedure to the completion of the procedure. The study timer was incorporated in the study IPAD and timing was performed by the nurse orchestrator.

SECONDARY OUTCOMES:
Effectiveness of the distraction technique | Twelve months
  Both patient groups assessed the effectiveness of their distraction techniques following the procedure by using a Visual analogue/FACES scale answering 3 anchored questions. 1) "Did the distraction technique keep you/your child /your patient engaged?" The anchors were 0=It really kept them engaged and 100=It really did not keep them engaged. 2) "Do you think the distraction technique/s changed you/your child/your patient's nervousness/anxiety level during the IV procedure?" The anchor of 0=it decreased nervousness/anxiety a lot, 100=it increased nervousness/anxiety a lot. 3) "How did the distraction technique/s affect pain during your/your child/your patient's IV procedure?" With 0=it made pain a lot better, 100=it made pain a lot worse.
Usability and Likeability | Twelve months
  For patients randomized to the VR arm, data on the use of the VR equipment was recorded by the nurse orchestrator at the end of each procedure. Data was categorized if the participant wore the VR equipment: 1) during the entire procedure, 2) part of the procedure or 3) only prior to the procedure. Participants were also asked to rate usability of the VR equipment, by using the VAS/FACES scale to answer "How easy was it for you/your child/your patient to use the VR equipment?" A score of 0 represented really easy to use and a score of 100 correlated with really hard to use. Lastly, participants were asked to use the VAS?FACES scale to answer a likeability question by "How much would you/your child/your patient like to use VR for future IV procedures?" A score of 0 equated to they would really like to use VR again and 100 meant they would really not like to use it again.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Dunn A, Patterson J, Biega CF, Grishchenko A, Luna J, Stanek JR, Strouse R. A Novel Clinician-Orchestrated Virtual Reality Platform for Distraction During Pediatric Intravenous Procedures in Children With Hemophilia: Randomized Controlled Trial. JMIR Serious Games. 2019 Jan 9;7(1):e10902. doi: 10.2196/10902. PMID 30626567